CLINICAL TRIAL: NCT02592772
Title: Manipulating Tobacco Constituents in Male Menthol Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HHC-2015-0128; 3R01DA036486-02S1 (NIH)
Record Dates: First submitted 2015-10-20; First posted 2015-10-30 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Nicotine Dependence
Keywords: menthol; nicotine; reduced nicotine; smoking; cigarette; cigarettes; men smoking; smoking research; nicotine dependence
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Reduced Nicotine Non-Menthol (RNC) (Experimental): Study participants will be randomized from their own brand of menthol cigarettes to the reduced nicotine non menthol cigarettes (RNC: NRC 200; 0.07 mg nicotine yield cigarettes without menthol) during the 6 week experimental phase.
  Interventions: Other: Reduced Nicotine Non-Menthol (RNC)
- Reduced Nicotine Menthol (RNC-Men) (Experimental): Study participants will be randomized from their own brand of menthol cigarettes to the reduced nicotine menthol cigarettes (RNC-Men: NRC 201; 0.07 mg reduced nicotine content menthol cigarettes) during the 6 week experimental phase.
  Interventions: Other: Reduced Nicotine Menthol (RNC-Men)
- Conventional Nicotine Non-Menthol (CN) (Experimental): Study participants will be randomized from their own brand of menthol cigarettes to the regular/conventional nicotine non menthol cigarettes (CN: NRC 600; 0.8 mg nicotine content) during the 6 week experimental phase.
  Interventions: Other: Conventional Nicotine Non-Menthol (CN)

INTERVENTIONS:
Other: Reduced Nicotine Non-Menthol (RNC) — Switch from own brand of cigarette to an investigational tobacco product with a reduced nicotine content of 0.07mg nicotine yield without menthol.
  Other Names: SPECTRUM Research Cigarette - NRC 200
  Arms: Reduced Nicotine Non-Menthol (RNC)
Other: Reduced Nicotine Menthol (RNC-Men) — Switch from own brand of cigarette to an investigational tobacco product with a reduced nicotine content of 0.07mg nicotine yield with menthol.
  Other Names: SPECTRUM Research Cigarette - NRC 201
  Arms: Reduced Nicotine Menthol (RNC-Men)
Other: Conventional Nicotine Non-Menthol (CN) — Switch from own brand of cigarette to an investigational tobacco product which contains conventional nicotine yield.
  Other Names: SPECTRUM Research Cigarette - NRC 600
  Arms: Conventional Nicotine Non-Menthol (CN)

SUMMARY:
This study examines the potential effect of reducing nicotine content or menthol or both in men. It will also examine whether there are gender differences in manipulating tobacco flavors and nicotine concentrations in cigarettes on smoking behavior.

DETAILED DESCRIPTION:
The FDA has the regulatory authority to reduce, but not eliminate, nicotine from cigarettes. The Tobacco Products Scientific Advisory Committee has noted, among other things, that removal of menthol cigarettes from the marketplace would benefit the public health. A parent study (NCT02048852) examines the potential impact of these two regulatory actions alone and in combination in female menthol smokers. This supplemental study will recruit an additional group of male menthol smokers, which will examine whether there are gender differences in manipulating flavors and nicotine concentrations in cigarettes on smoking behavior. The approach to add the opposite sex allows findings of sex/gender to be incorporated in the design and development of new technologies (i.e., modified cigarettes). Emerging research shows that women may be more responsive to the non-nicotine sensory aspects of smoking such as menthol flavor, whereas men may smoke primarily for nicotine intake. Consequently, this study expects to observe gender differences in response to manipulating flavors and nicotine content in cigarettes.

ELIGIBILITY:
Inclusion Criteria:

1. smoking at least 5 menthol cigarettes daily for the last year;
2. able to speak, read and understand English;
3. male age 18 -45 years of age;
4. stable residence;
5. not intending to quit smoking within the next 6 weeks.

Exclusion Criteria:

1. unstable psychiatric disorder (Psychiatric symptoms reported that cause current significant impairment in functioning or judgment such that the person's ability to come consistently for study appointments or render a decision regarding informed consent is in question.);
2. substance use which exceeds any of the following: marijuana use 3x/week, consuming 21 drinks/week or illicit drug use 1x/week;
3. history of cardiovascular disease;
4. current blood clot in arms or legs;
5. blood pressure >160/100;
6. unstable medical problems which may include but are not limited to immune system disorders, severe respiratory diseases, kidney or liver diseases, thyroid problems, substance abuse or dependence that would limit patients ability to follow experimental protocol
7. Serious quit attempts in the last 3 months;
8. regular use (e.g., greater than weekly) of tobacco products other than cigarettes;
9. currently using nicotine replacement or other tobacco cessation products

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Gender differences and change in number of investigational tobacco product(s) smoked per day as assessed by the Timeline Follow-Back (TLFB) | Baseline, 6 weeks, and 12 weeks
  Data analyses will include subjects from this study matched to female subjects from the parent study.

SECONDARY OUTCOMES:
Gender differences and changes in craving as assessed by Minnesota Nicotine Withdrawal Scale (MNWS). | Baseline, 6 weeks, and 12 weeks
Gender differences and changes in nicotine dependence as assessed by the Wisconsin Index of Smoking Dependence Motives (WISDM). | Baseline, 6 weeks, and 12 weeks
Gender differences and changes in nicotine dependence as assessed by the Fagerstrom Test of Nicotine Dependence (FTND) | Baseline, 6 weeks, and 12 weeks
Supertaster status as measured by genotyping for taster-receptor genes associated with taste behaviors. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Oncken, MD, MPH, Principal Investigator — UConn Health; Ellen Dornelas, PhD, Principal Investigator — Hartford HealthCare
Locations (2):
- United States (2):
  - UCONN Health Center, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut

IPD SHARING:
Plan to Share IPD: No